CLINICAL TRIAL: NCT02720068
Title: A Phase 1 Trial of MK-4280 as Monotherapy and in Combination With Pembrolizumab With or Without Chemotherapy or Lenvatinib (E7080/MK-7902) in Subjects With Advanced Solid Tumors
Brief Title: Study of Favezelimab (MK-4280) as Monotherapy and in Combination With Pembrolizumab (MK-3475) With or Without Chemotherapy or Lenvatinib (MK-7902) AND Favezelimab/Pembrolizumab (MK-4280A) as Monotherapy in Adults With Advanced Solid Tumors (MK-4280-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4280-001; MK-4280-001 (Other: Merck Protocol Number); 183971 (Other: JAPIC-CTI); 2017-001464-38 (EudraCT Number)
Record Dates: First submitted 2016-03-22; First posted 2016-03-25 (Estimated); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); Lymphocyte-activation gene 3 (LAG3, LAG-3, CD223)
MeSH Terms: conditions — Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; lenvatinib

STUDY DESIGN:
Intervention Model Description: Participants were allocated to arms in a non-random fashion, except in the case of those with gastric cancer enrolled in Part B, who were randomized 1:1 between Arm 2A and Arm 2B (favezelimab 200 mg and 800 mg, respectively). Part B initiated after determination of a favezelimab recommended phase 2 dose (RP2D) from Part A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Part A: Favezelimab 7 mg Monotherapy (Experimental): Participants received favezelimab 7 mg intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab
- Part A: Favezelimab 21 mg Monotherapy (Experimental): Participants received favezelimab 21 mg IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab
- Part A: Favezelimab 70 mg Monotherapy (Experimental): Participants received favezelimab 70 mg IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab
- Part A: Favezelimab 210 mg Monotherapy (Experimental): Participants received favezelimab 210 mg IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab
- Part A: Favezelimab 700 mg Monotherapy (Experimental): Participants received favezelimab 700 mg IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab
- Part A: Favezelimab 7 mg + Pembrolizumab 200 mg (Experimental): Participants received favezelimab 7 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab
- Part A: Favezelimab 21 mg + Pembrolizumab 200 mg (Experimental): Participants received favezelimab 21 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab
- Part A: Favezelimab 70 mg + Pembrolizumab 200 mg (Experimental): Participants received favezelimab 70 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab
- Part A: Favezelimab 210 mg + Pembrolizumab 200 mg (Experimental): Participants received favezelimab 210 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab
- Part A: Favezelimab 700 mg + Pembrolizumab 200 mg (Experimental): Participants received favezelimab 700 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab
- Part B: Favezelimab 800 mg Monotherapy (Arm 1) (Experimental): Participants received favezelimab 800 mg monotherapy IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab
- Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) (Experimental): Participants received favezelimab 200 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab
- Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) (Experimental): Participants received favezelimab 700 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab
- Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) (Experimental): Participants received favezelimab 800 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab
- Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) (Experimental): Participants received favezelimab 800 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle PLUS mFOLFOX7 (oxaliplatin 85 mg/m^2 IV, leucovorin [calcium folinate] 400 mg/m^2 IV, and fluorouracil [5-FU] 2400 mg/m^2 IV over 46 to 48 hours, every 2 weeks [Q2W]).
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab; Drug: Oxaliplatin; Drug: Leucovorin (Calcium Folinate); Drug: Fluorouracil [5-FU]
- Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) (Experimental): Participants received favezelimab 800 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle PLUS FOLFIRI (irinotecan 180 mg/m^2 IV, leucovorin [calcium folinate] 400 mg/m^2 IV and 5-FU 2400 mg/m^2 IV over 46 to 48 hours, Q2W).
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab; Drug: Irinotecan; Drug: Leucovorin (Calcium Folinate); Drug: Fluorouracil [5-FU]
- Part B: MK-4280A (Arm 5) (Experimental): Participants received MK-4280A, a coformulation of favezelimab 800 mg + pembrolizumab 200 mg IV infusion on Day 1 of each 21-day cycle.
  Interventions: Biological: Favezelimab/Pembrolizumab
- Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) (Experimental): Participants received favezelimab 800 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle PLUS oral lenvatinib 20 mg once daily.
  Interventions: Biological: Favezelimab; Biological: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Biological: Favezelimab — IV infusion
  Other Names: MK-4280
  Arms: Part A: Favezelimab 21 mg + Pembrolizumab 200 mg; Part A: Favezelimab 21 mg Monotherapy; Part A: Favezelimab 210 mg + Pembrolizumab 200 mg; Part A: Favezelimab 210 mg Monotherapy; Part A: Favezelimab 7 mg + Pembrolizumab 200 mg; Part A: Favezelimab 7 mg Monotherapy; Part A: Favezelimab 70 mg + Pembrolizumab 200 mg; Part A: Favezelimab 70 mg Monotherapy; Part A: Favezelimab 700 mg + Pembrolizumab 200 mg; Part A: Favezelimab 700 mg Monotherapy; Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A); Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3); Part B: Favezelimab 800 mg Monotherapy (Arm 1)
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Part A: Favezelimab 21 mg + Pembrolizumab 200 mg; Part A: Favezelimab 210 mg + Pembrolizumab 200 mg; Part A: Favezelimab 7 mg + Pembrolizumab 200 mg; Part A: Favezelimab 70 mg + Pembrolizumab 200 mg; Part A: Favezelimab 700 mg + Pembrolizumab 200 mg; Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A); Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3)
Drug: Oxaliplatin — IV infusion
  Other Names: ELOXATIN®
  Arms: Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3)
Drug: Irinotecan — IV infusion
  Other Names: CAMPTOSAR®
  Arms: Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4)
Drug: Leucovorin (Calcium Folinate) — IV infusion
  Other Names: WELLCOVORIN®
  Arms: Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3)
Drug: Fluorouracil [5-FU] — IV infusion
  Other Names: ADRUCIL®
  Arms: Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4); Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3)
Biological: Favezelimab/Pembrolizumab — IV infusion
  Other Names: MK-4280A
  Arms: Part B: MK-4280A (Arm 5)
Drug: Lenvatinib — Oral
  Other Names: E7080; MK-7902; LENVIMA®
  Arms: Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6)

SUMMARY:
This is a safety and pharmacokinetics study of favezelimab as monotherapy and in combination with pembrolizumab AND favezelimab/pembrolizumab as monotherapy in adults with metastatic solid tumors for which there is no available therapy which may convey clinical benefit. Part A of this study is a dose escalation design in which participants receive favezelimab as monotherapy or favezelimab in combination with pembrolizumab. Part B is a dose confirmation design to estimate the recommended Phase 2 dose (RP2D), as determined by dose-limiting toxicity, for favezelimab in combination with pembrolizumab or pembrolizumab and lenvatinib in participants with advanced solid tumors. Part B will also assess the efficacy of favezelimab as monotherapy; favezelimab in combination with pembrolizumab with and without chemotherapy; favezelimab in combination with pembrolizumab and lenvatinib; and favezelimab/pembrolizumab as monotherapy in expansion cohorts. Participants who have completed the initial course of treatment and have investigator-determined progressive disease may be eligible for a second course of an additional 17 cycles of study treatment.

DETAILED DESCRIPTION:
All participants who completed the first course were eligible for second course treatment after Sponsor consultation if there was investigator-determined progressive disease after initial treatment had been been completed.

ELIGIBILITY:
Inclusion Criteria:

* Part A and Part B: Has histologically or cytologically-confirmed metastatic solid tumor.
* Has measurable disease by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) 1.1 criteria.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrates adequate organ function.
* If female, is not pregnant or breastfeeding, and if of child-bearing potential, is willing to use an adequate method of contraception for the course of the study and for at least 180 days after the last dose of chemotherapy, 120 days after the last dose of pembrolizumab or favezelimab, or 30 days after the last dose of lenvatinib, whichever occurs last.
* If male with a female partner(s) of child-bearing potential, both must agree to use an adequate method of contraception starting with the first dose of study drug through 95 days after the last dose of study drug.

Exclusion Criteria:

* Has had chemotherapy, radiation or biological cancer therapy within 4 weeks prior to the first dose of study drug, or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 0 or 1 from the AEs due to cancer therapeutics administered more than 4 weeks earlier (this includes participants with previous immunomodulatory therapy with residual immune-related [ir]AEs).
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug.
* Has received previous treatment with another agent targeting the lymphocyte-activation gene 3 (LAG-3) receptor.
* Has received previous treatment with an immunomodulatory therapy (e.g., anti-programmed cell death-1/anti-programmed cell death-ligand 1 [anti-PD-1/anti-PD-L1] or cytotoxic T-lymphocyte-associated protein 4 [CTLA 4] agent) and was discontinued from that therapy due to a Grade 3 or higher irAE.
* Is expected to require any other form of antineoplastic therapy while on study.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy in excess of replacement doses, or on any other form of immunosuppressive medication.
* Has a history of a previous, additional malignancy, unless potentially curative treatment has been completed, with no evidence of malignancy for 5 years. Time frame exceptions include successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer or in situ cervical cancer, or other in situ cancers.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has had a severe hypersensitivity reaction to treatment with another monoclonal antibody.
* Has an active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy.
* Has an active infection requiring therapy.
* Has history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has had a prior stem cell or bone marrow transplant.
* Has a known history of or screens positive for Human Immunodeficiency Virus (HIV), active chronic or acute Hepatitis B or Hepatitis C.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Is a regular user as determined by investigator judgement (including "recreational use") of any illicit drugs or has a recent history (within the last year) of substance abuse (including alcohol), at the time of signing informed consent.
* Has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible.
* Has clinically significant heart disease that affects normal activities.
* Has received a live-virus vaccine within 30 days of planned start of study drug. Seasonal flu vaccines that do not contain live virus are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Background] Study of Favezelimab (MK-4280) as Monotherapy and in Combination With Pembrolizumab (MK-3475) With or Without Chemotherapy or Lenvatinib (MK-7902) AND Favezelimab/Pembrolizumab (MK-4280A) as Monotherapy in Adults With Advanced Solid Tumors (MK-4280-001) - Full Text View - ClinicalTrials.gov
- [Result] Garralda E, Sukari A, Lakhani NJ, Patnaik A, Lou Y, Im SA, Golan T, Geva R, Wermke M, de Miguel M, Palcza J, Jha S, Chaney M, Abraham AK, Healy J, Falchook GS. A first-in-human study of the anti-LAG-3 antibody favezelimab plus pembrolizumab in previously treated, advanced microsatellite stable colorectal cancer. ESMO Open. 2022 Dec;7(6):100639. doi: 10.1016/j.esmoop.2022.100639. Epub 2022 Dec 6. PMID 36493599
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant received 2 randomization numbers due to an erroneous initial randomization, but is only counted once in Participant Flow due to the rapid correction and drug administration only happening after the correction.
Groups:
- Part B: Favezelimab 800 mg Monotherapy (Arm 1): Participants received favezelimab 800 mg monotherapy IV infusion on Day 1 of each 21-day cycle. 9 participants with confirmed disease progression per irRECIST 1.1 switched over to Arm 2C and received favezelimab 800 mg + pembrolizumab 200 mg on Day 1 of each 21-day cycle for up to 35 cycles. Any events occurring after that switch-over are reported in a separate arm instead of this one.
Period: Overall Study
Arm/Group | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 700 mg Monotherapy | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: MK-4280A (Arm 5) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6)
Started | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 21 | 206 | 40 | 41 | 59 | 20 | 21 | 40
Treated | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 20 | 205 | 40 | 41 | 58 | 20 | 20 | 40
Switched Over to Favezelimab + Pembrolizumab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Second Course of Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 21 | 206 | 40 | 41 | 59 | 20 | 21 | 40
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 3 | 2 | 1 | 2 | 1 | 2 | 2 | 3 | 1 | 20 | 166 | 34 | 30 | 45 | 16 | 20 | 28
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive Disease | 2 | 3 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 2 | 4 | 4 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 27 | 2 | 8 | 7 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 700 mg Monotherapy | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: MK-4280A (Arm 5) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 21 | 206 | 40 | 41 | 59 | 20 | 21 | 40 | 481
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (15.5) | 59.3 (10.1) | 68.7 (15.3) | 48.7 (6.1) | 52.0 (14.7) | 54.0 (12.2) | 52.3 (17.1) | 64.7 (7.5) | 55.3 (12.4) | 68.7 (9.6) | 60.3 (10.6) | 58.1 (11.2) | 58.5 (12.0) | 57.9 (10.9) | 56.3 (9.7) | 58.3 (12.1) | 59.5 (9.9) | 61.1 (11.0) | 58.3 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 2 | 1 | 1 | 1 | 2 | 2 | 1 | 11 | 73 | 15 | 17 | 11 | 5 | 9 | 21 | 180
  Male | 1 | 2 | 1 | 1 | 2 | 2 | 2 | 1 | 1 | 2 | 10 | 133 | 25 | 24 | 48 | 15 | 12 | 19 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 25 | 6 | 8 | 4 | 1 | 7 | 1 | 58
  Not Hispanic or Latino | 2 | 5 | 3 | 3 | 3 | 2 | 2 | 2 | 3 | 1 | 19 | 174 | 33 | 32 | 52 | 19 | 12 | 39 | 406
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 1 | 1 | 3 | 0 | 2 | 0 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 36 | 11 | 9 | 20 | 7 | 2 | 12 | 98
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 1 | 3 | 1 | 2 | 0 | 15
  White | 1 | 6 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 19 | 164 | 29 | 31 | 30 | 12 | 17 | 25 | 356
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: DLTs were assessed during the first cycle (21 days) & were defined as: Grade (Gr) 4 nonhematologic toxicity; Gr 4 hematologic toxicity lasting ≥7 days, except Gr 4 thrombocytopenia of any duration or Gr 3 thrombocytopenia associated with bleeding; Gr 3 nonhematologic toxicity lasting ≥3 days despite optimal supportive care (with exceptions); Gr 3 or 4 nonhematologic lab abnormality (if medical intervention was required, lead to hospitalization, or persisted for >1 week); Gr 3 or 4 febrile neutropenia; any drug-related AE that caused the participant to discontinue treatment during Cycle 1; Grade 5 toxicity; Any treatment-related toxicity that causes ≥2-week delay in initiation of Cycle 2.
Time Frame: Up to 21 days (Cycle 1)
Population: All participants who received ≥1 dose of study treatment prior to determination of maximum tolerated dose, and were observed for safety for 21 days after their first dose of assigned treatment or experienced a DLT prior to 21 days after their first dose of assigned treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Favezelimab 700 mg Monotherapy: Participants received favezelimab 710 mg IV infusion on Day 1 of each 21-day cycle.
Arm/Group | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 700 mg Monotherapy | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: MK-4280A (Arm 5) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6)
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 19 | 198 | 38 | 38 | 20 | 20 | 38 | 39
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 31.3 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A): Participants received favezelimab 200 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle. One participant received a second course for up to 17 cycles; any events occurring after initiating the second course were reported in a separate arm instead of this one.
- Part B: Favezelimab Switch Over to Favezelimab 800 mg + Pembrolizumab 200 mg (Switch Over to Arm 2C): Part B favezelimab monotherapy-treated participants (Arm 1) with confirmed disease progression per irRECIST 1.1 were allowed to switch over to Arm 2C and receive favezelimab 800 mg + pembrolizumab 200 mg on Day 1 of each 21-day cycle for up to 35 cycles.
- Part B: Second Course Favezelimab 200 mg + Pembrolizumab 200 mg (Second Course Arm 2A): One participant enrolled in Arm 2A received a second course of favezelimab 200 mg + Pembrolizumab 200 mg on Day 1 of each 21-day cycle for up to 17 cycles.
Arm/Group | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 700 mg Monotherapy | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: MK-4280A (Arm 5) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab Switch Over to Favezelimab 800 mg + Pembrolizumab 200 mg (Switch Over to Arm 2C) | Part B: Second Course Favezelimab 200 mg + Pembrolizumab 200 mg (Second Course Arm 2A)
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 20 | 205 | 40 | 41 | 20 | 20 | 58 | 40 | 9 | 1
Participants | 3 | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 19 | 196 | 40 | 41 | 20 | 20 | 55 | 40 | 7 | 1

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 28.3 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 700 mg Monotherapy | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: MK-4280A (Arm 5) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab Switch Over to Favezelimab 800 mg + Pembrolizumab 200 mg (Switch Over to Arm 2C) | Part B: Second Course Favezelimab 200 mg + Pembrolizumab 200 mg (Second Course Arm 2A)
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 20 | 205 | 40 | 41 | 20 | 20 | 58 | 40 | 9 | 1
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 22 | 5 | 2 | 6 | 0 | 5 | 11 | 1 | 0

4. Secondary Outcome: Objective Response Rate (ORR) for Part B Participants
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experienced a CR or PR is presented.
Time Frame: Up to approximately 92 months
Population: All participants enrolled in Part B with a baseline scan with measurable disease by investigator assessment, who received ≥1 dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Colorectal Cancer Participants in Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A): Participants with colorectal cancer received favezelimab 200 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
- HNSCC Participants in Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A): Participants with head and neck squamous cell cancer (HNSCC) received favezelimab 200 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
- Gastric Cancer Participants in Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A): Participants with gastric cancer received favezelimab 200 mg IV infusion on Day 1 of each 21-day cycle PLUS pembrolizumab 200 mg IV infusion administered sequentially on Day 1 of each 21-day cycle.
- Colorectal Cancer Participants in Part B: MK-4280A (Arm 5): Participants with colorectal cancer received MK-4280A, a coformulation of favezelimab 800 mg + pembrolizumab 200 mg IV infusion on Day 1 of each 21-day cycle.
- China Enrollment in Part B: MK-4280A (Arm 5): Participants enrolled in China received MK-4280A, a coformulation of favezelimab 800 mg + pembrolizumab 200 mg IV infusion on Day 1 of each 21-day cycle.
Arm/Group | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Colorectal Cancer Participants in Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | HNSCC Participants in Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Gastric Cancer Participants in Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Colorectal Cancer Participants in Part B: MK-4280A (Arm 5) | China Enrollment in Part B: MK-4280A (Arm 5) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6)
Number analyzed (Participants) | 20 | 105 | 60 | 40 | 40 | 41 | 39 | 19 | 20 | 20 | 40
Percentage of Participants | 0.0 [0.0 to 16.8] | 3.8 [1.0 to 9.5] | 15.0 [7.1 to 26.6] | 7.5 [1.6 to 20.4] | 15.0 [5.7 to 29.8] | 7.3 [1.5 to 19.9] | 5.1 [0.6 to 17.3] | 10.5 [1.3 to 33.1] | 25.0 [8.7 to 49.1] | 0.0 [0.0 to 16.8] | 7.5 [1.6 to 20.4]
Statistical Analysis 1: Comparison: Gastric Cancer Participants in Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) vs Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B); Test type: Other — Difference in Percentage; Mean Difference (Final Values) = 7.5, 95% CI 2-sided [-7.3 to 22.9] — Confidence interval based on Miettinen & Nurminen method

5. Secondary Outcome: Area Under the Curve From Time 0 to Infinity (AUC0-inf) of Favezelimab
Description: Blood for serum samples was collected at pre-specified time points to determine the AUC0-inf of favezelimab. In addition to time points listed in Time Frame, participants enrolled in mainland China also had samples drawn predose on Day 1 of Cycle 5 and postdose on Day 2 of Cycles 4 and 8. Per protocol, different arms had different sampling schedules and therefore were not analyzed for all cycles.
Time Frame: Predose, 2 hours post start of infusion, and post infusion on Day 1 of cycles 1-4 and 8; Day 2 postdose in cycle 1; Days 8 and 15 in cycles 2, 4, and 8; and at the discontinuation and safety follow-up visit if performed prior to the end of Cycle 8
Population: All participants who complied with the protocol sufficiently to ensure that generated data likely exhibiting the effects of treatment, according to the underlying scientific model
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*μg/mL
Groups:
- Pooled Favezelimab 7 mg: This arm is a protocol-specified pooled arm of all participants who received favezelimab 7 mg intravenous (IV) infusion on Day 1 of each 21-day cycle.
- Pooled Favezelimab 21 mg: This arm is a protocol-specified pooled arm of all participants who received favezelimab 21 mg IV infusion on Day 1 of each 21-day cycle.
- Pooled Favezelimab 70 mg: This arm is a protocol-specified pooled arm of all participants who received favezelimab 70 mg IV infusion on Day 1 of each 21-day cycle.
- Pooled Favezelimab 200 mg: This arm is a protocol-specified pooled arm of all participants who received favezelimab 200 mg IV infusion on Day 1 of each 21-day cycle.
- Pooled Favezelimab 210 mg: This arm is a protocol-specified pooled arm of all participants who received favezelimab 210 mg IV infusion on Day 1 of each 21-day cycle.
- Pooled Favezelimab 700 mg: This arm is a protocol-specified pooled arm of all participants who received favezelimab 700 mg IV infusion on Day 1 of each 21-day cycle.
- Pooled Favezelimab 800 mg: This arm is a protocol-specified pooled arm of all participants who received favezelimab 800 mg IV infusion on Day 1 of each 21-day cycle, including participants who received it as part of a coformulation with pembrolizumab (MK-4280A).
Arm/Group | Pooled Favezelimab 7 mg | Pooled Favezelimab 21 mg | Pooled Favezelimab 70 mg | Pooled Favezelimab 200 mg | Pooled Favezelimab 210 mg | Pooled Favezelimab 700 mg | Pooled Favezelimab 800 mg | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 700 mg Monotherapy | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: MK-4280A (Arm 5)
Number analyzed (Participants) | 6 | 7 | 6 | 187 | 6 | 45 | 184 | 3 | 6 | 3 | 3 | 3 | 18 | 3 | 2 | 3 | 188 | 3 | 3 | 40 | 40 | 20 | 33 | 20 | 54
Day*μg/mL
  Cycle 1: number analyzed (Participants) | 6 | 7 | 6 | 187 | 6 | 45 | 184 | 3 | 6 | 3 | 3 | 3 | 18 | 3 | 1 | 3 | 188 | 3 | 3 | 40 | 40 | 20 | 33 | 20 | 54
  Cycle 1 | 7.12 (58.8) | 34.6 (45.4) | 98.8 (42.7) | 305 (48.4) | 365 (39.8) | 1480 (39.6) | 1620 (54.7) | 10.5 (49) | 37.4 (43.3) | 99.3 (28.6) | 341 (51) | 1590 (21.5) | 1820 (46.6) | 4.81 (25.7) | 21.5 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 98.3 (63.7) | 305 (48.3) | 391 (36.1) | 1610 (36.5) | 1440 (41.6) | 1430 (46.4) | 1670 (40.3) | 1870 (75.1) | 2010 (54.5) | 1430 (49.6)
  Cycle 2: number analyzed (Participants) | 4 | 6 | 6 | 123 | 6 | 36 | 113 | 1 | 6 | 3 | 3 | 3 | 10 | 3 | 0 | 3 | 127 | 3 | 3 | 30 | 25 | 17 | 0 | 19 | 44
  Cycle 2 | 8.28 (45.8) | 33.1 (41.3) | 56.0 (179.4) | 330 (58.1) | 335 (48.5) | 1730 (53.1) | 1850 (59.2) | 14.6 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 33.1 (41.3) | 60.0 (92.4) | 298 (51.6) | 1640 (20.5) | 2200 (42.8) | 6.86 (27.3) |  | 52.2 (429.4) | 324 (58.7) | 378 (53.1) | 2330 (18.4) | 1690 (57.4) | 1450 (49.9) | 2300 (46.6) |  | 2690 (55) | 1580 (61.9)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 3 |  |  |  | 248 (33.6) |  | 2000 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 3880 (16.9) |  |  |  |  |  | 3880 (16.8) |  |  |  | 248 (33.6) |  |  | 2000 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant |  |  |  |  |
  Cycle 4: number analyzed (Participants) | 3 | 2 | 3 | 44 | 3 | 13 | 37 | 0 | 0 | 1 | 2 | 0 | 4 | 3 | 2 | 2 | 45 | 1 | 1 | 12 | 6 | 5 | 0 | 3 | 19
  Cycle 4 | 9.38 (22.3) | 13.7 (79.5) | 88.2 (80.4) | 329 (71.5) | 166 (114.5) | 1870 (56.5) | 1860 (58.6) |  |  | 46.1 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 113 (109.9) |  | 2880 (55.2) | 9.38 (22.3) | 13.7 (79.5) | 122 (66.4) | 330 (70.6) | 357 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 1240 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 1940 (57.5) | 1570 (40.7) | 2370 (44.6) |  | 2070 (73.8) | 1640 (62.4)
  Cycle 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Cycle 8 |  |  |  |  |  |  | 2030 (67.6) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 2030 (67.6)

6. Secondary Outcome: Area Under the Curve From Time 0 to 21 Days (AUC0-21 Days) of Favezelimab
Description: Blood for serum samples was collected at pre-specified time points to determine the AUC0-21 Days of favezelimab. In addition to time points listed in Time Frame, participants enrolled in mainland China also had samples drawn predose on Day 1 of Cycle 5 and postdose on Day 2 of Cycles 4 and 8. Per protocol, different arms had different sampling schedules and therefore were not analyzed for all cycles.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*μg/mL
Arm/Group | Pooled Favezelimab 7 mg | Pooled Favezelimab 21 mg | Pooled Favezelimab 70 mg | Pooled Favezelimab 200 mg | Pooled Favezelimab 210 mg | Pooled Favezelimab 700 mg | Pooled Favezelimab 800 mg | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 700 mg Monotherapy | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: MK-4280A (Arm 5)
Number analyzed (Participants) | 6 | 9 | 6 | 191 | 6 | 46 | 188 | 3 | 6 | 3 | 3 | 3 | 18 | 3 | 3 | 3 | 191 | 3 | 3 | 40 | 40 | 20 | 36 | 20 | 58
Day*μg/mL
  Cycle 1 | 7.29 (58.4) | 37.5 (41.1) | 96.1 (39.6) | 285 (42.8) | 353 (38.4) | 1300 (34.1) | 1430 (48.1) | 11.0 (38.6) | 36.5 (42.4) | 97.2 (28.5) | 333 (49.6) | 1440 (23.2) | 1550 (35.8) | 4.82 (28.5) | 39.6 (47.7) | 95.0 (57.5) | 285 (42.8) | 374 (34.9) | 1370 (30.0) | 1290 (35.5) | 1330 (40.5) | 1420 (34.8) | 1640 (71.9) | 1630 (41.6) | 1290 (43.7)
  Cycle 2: number analyzed (Participants) | 5 | 6 | 6 | 133 | 6 | 36 | 120 | 2 | 6 | 3 | 3 | 3 | 12 | 3 | 0 | 3 | 133 | 3 | 3 | 30 | 27 | 17 | 0 | 20 | 44
  Cycle 2 | 7.83 (73.1) | 32.7 (40.1) | 56.4 (154.4) | 300 (51.4) | 321 (44.9) | 1480 (43) | 1570 (54.9) | 9.32 (184.6) | 32.7 (40.1) | 59.3 (88.6) | 292 (48.3) | 1470 (15.7) | 2140 (40.9) | 6.97 (25.7) |  | 53.7 (327.1) | 300 (51.4) | 353 (49.8) | 1640 (38.7) | 1460 (46) | 1260 (65.1) | 1820 (37.2) |  | 2050 (43.6) | 1400 (51.9)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 6 | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 6 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 3 |  |  |  | 241 (26.4) |  | 1770 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 2330 (51.5) |  |  |  |  |  | 2330 (51.5) |  |  |  | 241 (26.4) |  |  | 1770 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant |  |  |  |  |
  Cycle 4: number analyzed (Participants) | 3 | 2 | 3 | 45 | 3 | 13 | 37 | 0 | 0 | 1 | 2 | 0 | 4 | 3 | 2 | 2 | 45 | 1 | 1 | 12 | 6 | 5 | 0 | 4 | 19
  Cycle 4 | 9.57 (21.9) | 13.8 (81) | 89.6 (65) | 306 (63.4) | 174 (91) | 1620 (44.2) | 1710 (53.6) |  |  | 53.1 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 124 (83.4) |  | 2320 (34.6) | 9.57 (21.9) | 13.8 (81) | 116 (58.6) | 306 (63.4) | 341 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 1120 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 1670 (44.6) | 1500 (37.7) | 2070 (40.4) |  | 2330 (90.1) | 1490 (53.7)
  Cycle 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Cycle 8 |  |  |  |  |  |  | 1730 (51.8) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1730 (51.8)

7. Secondary Outcome: Maximum Serum Concentration (Cmax) of Favezelimab
Description: Blood for serum samples was collected at pre-specified time points to determine the Cmax of favezelimab. In addition to time points listed in Time Frame, participants enrolled in mainland China also had samples drawn predose on Day 1 of Cycle 5 and postdose on Day 2 of Cycles 4 and 8. Per protocol, different arms had different sampling schedules and therefore were not analyzed for all cycles.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Pooled Favezelimab 7 mg | Pooled Favezelimab 21 mg | Pooled Favezelimab 70 mg | Pooled Favezelimab 200 mg | Pooled Favezelimab 210 mg | Pooled Favezelimab 700 mg | Pooled Favezelimab 800 mg | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 700 mg Monotherapy | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: MK-4280A (Arm 5)
Number analyzed (Participants) | 6 | 9 | 6 | 203 | 6 | 46 | 195 | 3 | 6 | 3 | 3 | 3 | 18 | 3 | 3 | 3 | 203 | 3 | 3 | 40 | 41 | 20 | 38 | 20 | 58
μg/mL
  Cycle 1 | 2.39 (44.4) | 8.00 (22) | 21.9 (34.5) | 56.7 (32.2) | 77.4 (29.9) | 224 (27) | 248 (27.8) | 3.16 (44.9) | 8.62 (17.6) | 23.7 (21.9) | 74.9 (28.8) | 216 (19.9) | 271 (20.7) | 1.80 (17.9) | 6.88 (25.2) | 20.2 (48.9) | 56.7 (32.2) | 80.0 (37.5) | 252 (46.6) | 223 (26.5) | 248 (20.5) | 219 (23.6) | 281 (35.7) | 244 (33.9) | 234 (24.5)
  Cycle 2: number analyzed (Participants) | 5 | 9 | 6 | 163 | 6 | 40 | 138 | 2 | 6 | 3 | 3 | 3 | 15 | 3 | 3 | 3 | 163 | 3 | 3 | 34 | 35 | 18 | 0 | 20 | 50
  Cycle 2 | 2.44 (46.5) | 8.62 (29.2) | 19.3 (47.1) | 56.8 (34.9) | 76.7 (21.1) | 247 (32) | 247 (36.6) | 2.67 (97.4) | 9.65 (19.6) | 20.8 (21.8) | 70.6 (23.3) | 222 (15.8) | 301 (18) | 2.30 (21.4) | 6.88 (35.3) | 17.9 (74) | 56.8 (34.9) | 83.3 (19.2) | 238 (58.9) | 250 (31.5) | 228 (53.8) | 245 (25.5) |  | 266 (35.4) | 240 (28.6)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0 | 3 | 10 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 15 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Cycle 3 |  |  |  | 19.2 (138.4) |  | 150 (54) | 272 (45.6) |  |  |  |  |  | 272 (45.6) |  |  |  | 19.2 (138.4) |  |  | 150 (54) |  |  |  |  |
  Cycle 4: number analyzed (Participants) | 3 | 2 | 3 | 85 | 3 | 21 | 79 | 0 | 0 | 1 | 2 | 0 | 9 | 3 | 2 | 2 | 85 | 1 | 2 | 19 | 19 | 12 | 0 | 15 | 24
  Cycle 4 | 3.02 (6.2) | 6.11 (39.4) | 27.0 (30.6) | 58.6 (34.6) | 54.0 (9.3) | 253 (35) | 265 (32.2) |  |  | 24.5 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 55.3 (11.8) |  | 332 (19.4) | 3.02 (6.3) | 6.11 (39.4) | 28.3 (42.5) | 58.6 (34.6) | 51.4 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 145 (37.5) | 269 (29.4) | 252 (26.1) | 267 (35.7) |  | 262 (34.5) | 254 (35.9)
  Cycle 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Cycle 8 |  |  |  |  |  |  | 292 (26.6) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 292 (26.6)

8. Secondary Outcome: AUC0-inf of Pembrolizumab
Description: Blood for serum samples was collected at pre-specified time points to determine the AUC0-inf of pembrolizumab. In addition to time points listed in Time Frame, participants enrolled in mainland China also had samples drawn predose on Day 1 of Cycle 5 and postdose on Day 2 of Cycles 4 and 8. Per protocol, different arms had different sampling schedules and therefore were not analyzed for all cycles.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*μg/mL
Groups:
- Pooled Pembrolizumab 200 mg: This arm is a protocol-specified pooled arm of all participants who received pembrolizumab 200 mg intravenous (IV) infusion on Day 1 of each 21-day cycle, including participants who received it as part of a coformulation with favezelimab (MK-4280A).
Arm/Group | Pooled Pembrolizumab 200 mg | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: MK-4280A (Arm 5)
Number analyzed (Participants) | 412 | 3 | 2 | 3 | 197 | 3 | 3 | 40 | 40 | 20 | 36 | 20 | 54
Day*μg/mL
  Cycle 1: number analyzed (Participants) | 412 | 3 | 1 | 3 | 197 | 3 | 3 | 40 | 40 | 20 | 36 | 20 | 54
  Cycle 1 | 586 (38.9) | 662 (20.7) | 332 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 612 (40.8) | 564 (40.8) | 821 (18.2) | 543 (27.4) | 586 (39.1) | 589 (34.4) | 626 (26.7) | 623 (44.6) | 661 (32.9) | 619 (41.3)
  Cycle 2: number analyzed (Participants) | 292 | 3 | 2 | 3 | 150 | 3 | 3 | 32 | 30 | 18 | 0 | 19 | 45
  Cycle 2 | 843 (52.1) | 1060 (22.4) | 613 (100.5) | 940 (46.3) | 807 (50.6) | 727 (67.2) | 847 (23.2) | 877 (53.7) | 812 (41.4) | 1150 (59.8) |  | 1100 (48.8) | 861 (75.4)
  Cycle 3: number analyzed (Participants) | 5 | 0 | 0 | 0 | 7 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 3 | 846 (98) |  |  |  | 878 (72.1) |  |  | 1990 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant |  |  |  |  |
  Cycle 4: number analyzed (Participants) | 136 | 3 | 2 | 3 | 71 | 1 | 2 | 16 | 10 | 7 | 0 | 10 | 17
  Cycle 4 | 903 (49.2) | 1190 (17) | 503 (101.3) | 3650 (181.2) | 894 (47.9) | 962 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 528 (43.0) | 997 (56.6) | 848 (37.8) | 1000 (21.6) |  | 929 (35.7) | 1040 (73)
  Cycle 8: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Cycle 8 | 1980 (54.8) |  |  |  |  |  |  |  |  |  |  |  | 1970 (55)

9. Secondary Outcome: AUC0-21 Days of Pembrolizumab
Description: Blood for serum samples was collected at pre-specified time points to determine the AUC0-21 Days of pembrolizumab. In addition to time points listed in Time Frame, participants enrolled in mainland China also had samples drawn predose on Day 1 of Cycle 5 and postdose on Day 2 of Cycles 4 and 8. Per protocol, different arms had different sampling schedules and therefore were not analyzed for all cycles.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*μg/mL
Arm/Group | Pooled Pembrolizumab 200 mg | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: MK-4280A (Arm 5)
Number analyzed (Participants) | 424 | 3 | 3 | 3 | 197 | 3 | 3 | 40 | 40 | 20 | 38 | 20 | 54
Day*μg/mL
  Cycle 1 | 427 (31.5) | 418 (13) | 485 (49) | 382 (36.7) | 412 (31.1) | 556 (15.2) | 410 (30.0) | 422 (28.5) | 427 (25.2) | 431 (24) | 489 (39.3) | 447 (32.8) | 427 (34.2)
  Cycle 2: number analyzed (Participants) | 310 | 3 | 2 | 3 | 150 | 3 | 3 | 32 | 31 | 18 | 0 | 20 | 45
  Cycle 2 | 561 (38) | 615 (16.8) | 504 (88.8) | 597 (38.3) | 545 (36.6) | 662 (57.6) | 487 (27.9) | 588 (35.4) | 553 (25.1) | 618 (22.9) |  | 621 (32.4) | 547 (56.9)
  Cycle 3: number analyzed (Participants) | 13 | 0 | 0 | 0 | 11 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Cycle 3 | 543 (38.7) |  |  |  | 537 (40.1) |  |  | 577 (43.9) |  |  |  |  |
  Cycle 4: number analyzed (Participants) | 143 | 3 | 2 | 3 | 71 | 1 | 2 | 16 | 10 | 7 | 0 | 10 | 17
  Cycle 4 | 692 (39.3) | 805 (5) | 403 (74.6) | 1050 (79.9) | 670 (36.4) | 701 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 416 (15.7) | 754 (45.4) | 664 (31.9) | 769 (21.3) |  | 727 (36.7) | 705 (45.7)
  Cycle 8: number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Cycle 8 | 1040 (37.5) |  |  |  |  |  |  |  |  |  |  |  | 1040 (37.5)

10. Secondary Outcome: Cmax of Pembrolizumab
Description: Blood for serum samples was collected at pre-specified time points to determine the Cmax of pembrolizumab. In addition to time points listed in Time Frame, participants enrolled in mainland China also had samples drawn predose on Day 1 of Cycle 5 and postdose on Day 2 of Cycles 4 and 8. Per protocol, different arms had different sampling schedules and therefore were not analyzed for all cycles.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Pooled Pembrolizumab 200 mg | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: MK-4280A (Arm 5)
Number analyzed (Participants) | 435 | 3 | 3 | 3 | 204 | 3 | 3 | 40 | 41 | 20 | 38 | 20 | 57
μg/mL
  Cycle 1 | 59.6 (29.6) | 58.5 (14.9) | 60.0 (22.1) | 52.8 (51.5) | 58.7 (32.3) | 74.2 (39.1) | 57.4 (32.8) | 63.9 (26.2) | 61.3 (19.2) | 55.5 (20.5) | 65.0 (34) | 59.6 (30.9) | 56.6 (25.6)
  Cycle 2: number analyzed (Participants) | 338 | 3 | 3 | 3 | 165 | 3 | 3 | 34 | 35 | 18 | 0 | 20 | 51
  Cycle 2 | 67.5 (34.3) | 65.6 (21.2) | 78.7 (48.1) | 69.9 (37.1) | 66.7 (29.7) | 91.9 (14.1) | 67.6 (9.36) | 77.4 (33.7) | 67.0 (22.2) | 69.0 (22.6) |  | 69.9 (32.9) | 61.1 (55.1)
  Cycle 3: number analyzed (Participants) | 19 | 0 | 0 | 0 | 16 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
  Cycle 3 | 36.4 (41.9) |  |  |  | 36.7 (44.2) |  |  | 35.1 (35.3) |  |  |  |  |
  Cycle 4: number analyzed (Participants) | 186 | 3 | 2 | 3 | 86 | 1 | 2 | 19 | 19 | 12 | 0 | 15 | 24
  Cycle 4 | 76.1 (30.2) | 79.6 (7.8) | 59.3 (50.1) | 83.7 (83) | 75.3 (26.6) | 61.2 (NA) — NA= The Geometric Coefficient of Variation cannot be calculated for a single participant | 56.9 (3.48) | 90.7 (34.5) | 75.1 (25.1) | 76.0 (28.7) |  | 73.4 (27.3) | 74.1 (37.4)
  Cycle 8: number analyzed (Participants) | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Cycle 8 | 93.8 (25.8) |  |  |  |  |  |  |  |  |  |  |  | 93.8 (25.8)

11. Secondary Outcome: Predose Serum Concentration of Favezelimab
Description: Blood for serum samples was collected at pre-specified time points to determine the predose serum concentration of favezelimab, which is presented.
Time Frame: Predose on Day 1 of cycles 1-4, 6, and 8. Per protocol, different arms had different sampling schedules and therefore were not analyzed for all cycles.
Population: as for outcome 5
Measure: Median (Full Range); unit: μg/mL
Arm/Group | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg Monotherapy | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: MK-4280A (Arm 5)
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3 | 3 | 195 | 3 | 3 | 3 | 3 | 39 | 18 | 41 | 20 | 36 | 20 | 57
μg/mL
  Cycle 1 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Cycle 2: number analyzed (Participants) | 2 | 3 | 6 | 3 | 3 | 3 | 167 | 3 | 3 | 3 | 2 | 33 | 17 | 35 | 18 | 32 | 20 | 52
  Cycle 2 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.0361 [0.00 to 0.250] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.458] | 0.00 [0.00 to 1.87] | 1.52 [0.00 to 16.0] | 1.26 [0.361 to 2.24] | 3.28 [0.577 to 3.69] | 12.9 [11.7 to 20.7] | 23.6 [20.0 to 27.1] | 15.0 [1.62 to 50.0] | 21.8 [0.00 to 53.5] | 13.3 [0.00 to 45.1] | 25.2 [0.685 to 59.1] | 20.1 [0.00 to 62.7] | 27.0 [3.47 to 149] | 12.4 [0.00 to 58.1]
  Cycle 3: number analyzed (Participants) | 1 | 3 | 5 | 3 | 2 | 3 | 132 | 2 | 1 | 1 | 3 | 26 | 11 | 25 | 17 | 28 | 20 | 38
  Cycle 3 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.250] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 2.06] | 1.95 [0.00 to 29.9] | 0.225 [0.00 to 0.450] | 4.48 [4.48 to 4.48] | 28.2 [28.2 to 28.2] | 34.7 [32.3 to 36.8] | 23.7 [2.07 to 68.5] | 37.1 [3.31 to 389] | 14.8 [0.00 to 46.3] | 39.5 [3.81 to 81.3] | 35.8 [0.402 to 99.3] | 43.3 [6.34 to 119] | 19.1 [2.10 to 67.6]
  Cycle 4: number analyzed (Participants) | 0 | 3 | 0 | 2 | 1 | 2 | 91 | 2 | 1 | 0 | 2 | 19 | 10 | 19 | 13 | 24 | 15 | 23
  Cycle 4 |  | 0.00 [0.00 to 0.00] |  | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 1.09 [0.0559 to 2.12] | 2.26 [0.00 to 19.3] | 0.429 [0.00 to 0.858] | 4.54 [4.54 to 4.54] |  | 31.0 [27.4 to 34.5] | 25.0 [2.51 to 76.1] | 42.0 [4.43 to 78.4] | 20.5 [0.0659 to 60.9] | 45.6 [6.20 to 85.1] | 38.4 [0.00 to 164] | 51.2 [7.08 to 128] | 16.8 [1.06 to 68.5]
  Cycle 6: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 2 | 54 | 2 | 0 | 0 | 0 | 12 | 3 | 15 | 11 | 19 | 15 | 20
  Cycle 6 |  |  |  | 0.00 [0.00 to 0.00] | 15.1 [15.1 to 15.1] | 1.58 [0.0561 to 3.10] | 3.63 [0.00 to 19.2] | 50.6 [43.8 to 57.4] |  |  |  | 26.9 [6.53 to 113] | 35.1 [29.6 to 42.2] | 18.6 [0.729 to 68.4] | 40.3 [9.21 to 119] | 38.1 [1.14 to 119] | 59.6 [8.96 to 162] | 27.3 [0.464 to 246]
  Cycle 8: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2 | 31 | 1 | 0 | 0 | 0 | 6 | 2 | 7 | 11 | 13 | 8 | 15
  Cycle 8 |  | 0.00 [0.00 to 0.00] |  | 0.00 [0.00 to 0.00] |  | 1.09 [0.122 to 2.05] | 4.18 [0.00 to 13.7] | 0.00 [0.00 to 0.00] |  |  |  | 18.4 [9.48 to 113] | 30.8 [19.1 to 42.4] | 20.7 [5.62 to 35.9] | 51.1 [11.2 to 109] | 49.2 [1.48 to 161] | 64.3 [18.7 to 203] | 23.9 [0.289 to 84.8]

12. Secondary Outcome: AUC0-inf of Lenvatinib
Description: Blood for serum samples was collected at pre-specified time points to determine the AUC0-inf of lenvatinib.
Time Frame: Up to 4 hours postdose, and between 6-10 hours postdose on Cycle 1 Day 1; Predose and between 2-12 hours postdose on Cycle 1 Day 15; Predose, between 0.5-4 hours postdose, and between 6-10 hours postdose on Cycle 2 Day 1
Population: All participants who received ≥1 dose of lenvatinib and complied with the protocol sufficiently to ensure that generated data likely exhibiting the effects of treatment, according to the underlying scientific model
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ng/mL
Arm/Group | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6)
Number analyzed (Participants) | 35
Day*ng/mL
  Cycle 1 | NA (NA) — NA= AUC0-inf could not be calculated due to sparse data collection across participants
  Cycle 2: number analyzed (Participants) | 24
  Cycle 2 | NA (NA) — NA= AUC0-inf could not be calculated due to sparse data collection across participants

13. Secondary Outcome: AUC0-21 Days of Lenvatinib
Description: Blood for serum samples was collected at pre-specified time points to determine the AUC0-21 Days of lenvatinib.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*ng/mL
Arm/Group | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6)
Number analyzed (Participants) | 35
Day*ng/mL
  Cycle 1 | NA (NA) — NA= AUC0-21 Days could not be calculated due to sparse data collection across participants
  Cycle 2: number analyzed (Participants) | 24
  Cycle 2 | NA (NA) — NA= AUC0-21 Days could not be calculated due to sparse data collection across participants

14. Secondary Outcome: Cmax of Lenvatinib
Description: Blood for serum samples was collected at pre-specified time points to determine the Cmax of lenvatinib.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6)
Number analyzed (Participants) | 35
ng/mL
  Cycle 1 | NA (NA) — NA= Cmax Days could not be calculated due to sparse data collection across participants
  Cycle 2: number analyzed (Participants) | 24
  Cycle 2 | NA (NA) — NA= Cmax Days could not be calculated due to sparse data collection across participants

ADVERSE EVENTS:
Time Frame: Up to approximately 92 months
Description: AEs include all treated participants. Mortality includes all randomized participants. Per protocol, disease progression of cancer under study was not considered an AE unless hospitalization/death resulted, so "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" without hospitalization/death are excluded.
  Participants who received 2nd course/switch-over have AEs and mortality counted only in the arm corresponding to the latest treatment they received prior to the event
Arm/Group | Part A: Favezelimab 7 mg Monotherapy | Part A: Favezelimab 21 mg Monotherapy | Part A: Favezelimab 70 mg Monotherapy | Part A: Favezelimab 210 mg Monotherapy | Part A: Favezelimab 700 mg Monotherapy | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg | Part B: Favezelimab 800 mg Monotherapy (Arm 1) | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) | Part B: MK-4280A (Arm 5) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) | Part B: Favezelimab Switch Over to Favezelimab 800 mg + Pembrolizumab 200 mg (Switch Over to Arm 2C) | Part B: Second Course Favezelimab 200 mg + Pembrolizumab 200 mg (Second Course Arm 2A)
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/6 | 3/3 | 1/3 | 2/3 | 1/3 | 2/3 | 2/3 | 3/3 | 2/3 | 11/21 | 172/206 | 35/40 | 36/41 | 50/59 | 16/20 | 20/21 | 28/40 | 9/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/6 | 0/3 | 1/3 | 1/3 | 1/3 | 0/3 | 2/3 | 2/3 | 2/3 | 3/20 | 69/205 | 17/40 | 12/41 | 20/58 | 9/20 | 6/20 | 23/40 | 1/9 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 5/6 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 18/20 | 185/205 | 39/40 | 40/41 | 54/58 | 20/20 | 20/20 | 40/40 | 7/9 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Favezelimab 7 mg Monotherapy (N=3) | Part A: Favezelimab 21 mg Monotherapy (N=6) | Part A: Favezelimab 70 mg Monotherapy (N=3) | Part A: Favezelimab 210 mg Monotherapy (N=3) | Part A: Favezelimab 700 mg Monotherapy (N=3) | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg (N=3) | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg (N=3) | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg (N=3) | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg (N=3) | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg (N=3) | Part B: Favezelimab 800 mg Monotherapy (Arm 1) (N=20) | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) (N=205) | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) (N=40) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) (N=41) | Part B: MK-4280A (Arm 5) (N=58) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) (N=20) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) (N=20) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) (N=40) | Part B: Favezelimab Switch Over to Favezelimab 800 mg + Pembrolizumab 200 mg (Switch Over to Arm 2C) (N=9) | Part B: Second Course Favezelimab 200 mg + Pembrolizumab 200 mg (Second Course Arm 2A) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma prolapse (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Favezelimab 7 mg Monotherapy (N=3) | Part A: Favezelimab 21 mg Monotherapy (N=6) | Part A: Favezelimab 70 mg Monotherapy (N=3) | Part A: Favezelimab 210 mg Monotherapy (N=3) | Part A: Favezelimab 700 mg Monotherapy (N=3) | Part A: Favezelimab 7 mg + Pembrolizumab 200 mg (N=3) | Part A: Favezelimab 21 mg + Pembrolizumab 200 mg (N=3) | Part A: Favezelimab 70 mg + Pembrolizumab 200 mg (N=3) | Part A: Favezelimab 210 mg + Pembrolizumab 200 mg (N=3) | Part A: Favezelimab 700 mg + Pembrolizumab 200 mg (N=3) | Part B: Favezelimab 800 mg Monotherapy (Arm 1) (N=20) | Part B: Favezelimab 200 mg + Pembrolizumab 200 mg (Arm 2A) (N=205) | Part B: Favezelimab 700 mg + Pembrolizumab 200 mg (Arm 2B) (N=40) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg (Arm 2C) (N=41) | Part B: MK-4280A (Arm 5) (N=58) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + mFOLFOX7 (Arm 3) (N=20) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + FOLFIRI (Arm 4) (N=20) | Part B: Favezelimab 800 mg + Pembrolizumab 200 mg + Lenvatinib 20 mg (Arm 6) (N=40) | Part B: Favezelimab Switch Over to Favezelimab 800 mg + Pembrolizumab 200 mg (Switch Over to Arm 2C) (N=9) | Part B: Second Course Favezelimab 200 mg + Pembrolizumab 200 mg (Second Course Arm 2A) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 42 (49) | 8 (13) | 4 (4) | 9 (12) | 2 (2) | 3 (4) | 3 (3) | 1 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (18) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 8 (36) | 5 (7) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (7) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 15 (15) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 48 (50) | 7 (7) | 9 (9) | 8 (8) | 6 (6) | 1 (1) | 16 (17) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 26 (26) | 5 (5) | 5 (5) | 6 (6) | 3 (3) | 3 (3) | 7 (8) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (9) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 14 (14) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 24 (25) | 10 (10) | 7 (7) | 7 (7) | 8 (9) | 7 (10) | 8 (10) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 38 (50) | 8 (12) | 5 (5) | 9 (9) | 7 (14) | 11 (23) | 24 (45) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 2 (3) | 5 (5) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 6 (6) | 45 (51) | 15 (18) | 8 (8) | 8 (8) | 11 (29) | 12 (16) | 12 (19) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 5 (5) | 2 (3) | 4 (4) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 28 (32) | 7 (11) | 4 (5) | 5 (5) | 10 (15) | 11 (16) | 11 (19) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 26 (31) | 9 (11) | 6 (6) | 2 (2) | 4 (6) | 3 (5) | 9 (12) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 6 (7) | 59 (63) | 15 (15) | 11 (13) | 12 (13) | 11 (11) | 8 (12) | 11 (13) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (4) | 5 (6) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 12 (12) | 2 (3) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 38 (48) | 9 (17) | 7 (8) | 5 (6) | 6 (10) | 3 (4) | 5 (5) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (10) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 8 (12) | 4 (4) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 10 (20) | 0 (0) | 3 (4) | 2 (3) | 5 (10) | 3 (5) | 3 (3) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 16 (18) | 4 (4) | 9 (9) | 5 (5) | 6 (11) | 1 (1) | 8 (11) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 3 (10) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 23 (26) | 7 (8) | 9 (9) | 6 (6) | 8 (15) | 0 (0) | 9 (13) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 21 (23) | 7 (7) | 6 (6) | 6 (7) | 4 (9) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 8 (8) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 12 (13) | 4 (5) | 2 (2) | 3 (4) | 2 (3) | 1 (1) | 4 (7) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 18 (20) | 4 (4) | 6 (6) | 6 (6) | 5 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (15) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (6) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 7 (11) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 3 (6) | 1 (1) | 3 (5) | 3 (5) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (4) | 0 (0) | 1 (1) | 5 (14) | 7 (7) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 7 (39) | 1 (3) | 7 (9) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 8 (8) | 2 (2) | 5 (5) | 5 (5) | 6 (6) | 2 (2) | 7 (8) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 7 (33) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 42 (45) | 13 (19) | 7 (7) | 12 (12) | 7 (8) | 5 (8) | 11 (14) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 12 (17) | 3 (4) | 0 (0) | 8 (9) | 2 (2) | 4 (6) | 5 (6) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 2 (3) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 20 (26) | 6 (11) | 5 (5) | 9 (10) | 1 (1) | 4 (8) | 6 (6) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 17 (18) | 5 (5) | 3 (3) | 5 (7) | 4 (5) | 3 (8) | 2 (2) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 4 (4) | 6 (8) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 5 (6) | 4 (4) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 16 (17) | 5 (6) | 3 (4) | 5 (5) | 5 (7) | 4 (6) | 6 (6) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 7 (15) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 12 (13) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (22) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 27 (28) | 6 (9) | 10 (10) | 8 (8) | 4 (5) | 5 (6) | 6 (8) | 1 (1) | 0 (0)
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 16 (16) | 2 (2) | 8 (8) | 5 (5) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 21 (21) | 5 (5) | 5 (5) | 9 (13) | 2 (5) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 17 (19) | 5 (5) | 4 (5) | 8 (9) | 3 (4) | 5 (10) | 7 (7) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 27 (34) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 8 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT02720068/Prot_SAP_000.pdf